CLINICAL TRIAL: NCT05205421
Title: A Single-Arm, Open-Label, Exploratory Study to Evaluate Safety and Efficacy of Oncolytic Virus Injection (RT-01) in Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of Oncolytic Virus Injection (RT-01) in Patients With Extensive-Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Wang Zishu, Director of the Department of Medical Oncology, The First Affiliated Hospital of Bengbu Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LWY21076CBY2
Record Dates: First submitted 2022-01-19; First posted 2022-01-25 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumor
Keywords: RT-01; Oncolytic Virus; PD-L1 Inhibitor; immunotherapy; Intravenous Injection; Small-cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncolytic Virus Injection(RT-01) (Experimental): RT-01 will be administered by intravenously;
  Interventions: Biological: Oncolytic Virus Injection(RT-01)

INTERVENTIONS:
Biological: Oncolytic Virus Injection(RT-01) — Intravenous injection a single dose of RT-01

SUMMARY:
This is a single-arm, open-label, clinical pharmacology study to evaluate safety and efficacy of oncolytic virus injection(RT-01) in Patients With Extensive-Stage Small Cell Lung Cancer.

The purpose of this study is to evaluate the safety and tolerability, antitumor activity, The immunoreactivity, The immunogenicity, pharmacokinetics and virus shedding of RT-01.

DETAILED DESCRIPTION:
This is an investigator initiated , single-arm, open-label clinical pharmacology study of RT-01 as a single agent given via Intravenous injection in Patients With Extensive-Stage Small Cell Lung Cancer.

RT-01 will be administered as a single dose on day 1 in patients with advanced solid tumors. Durvalumab will be administered intravenously every 3 weeks starting on day 5 after RT-1 on day 1 for 4 cycles，then followed by every 4 weeks. This study is planned to enroll 10-20 patients with Extensive-Stage Small Cell Lung Cancer.

Considering the benefits of the subjects, the investigator deems that higher doses can be explored, then a higher-dose cohort will be carried out. The purpose of this study is to assess the safety and tolerability, antitumor activity, The immunoreactivity, The immunogenicity, pharmacokinetics and virus shedding of RT-01.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years;
* Subjects must have histologically or cytologically confirmed diagnosis of advanced solid tumor(s) who have failed in standard therapy (disease progression or intolerance) and no effective treatment, or have no standard therapy, or have failed to obtain standard treatment due to objective conditions ;
* Subjects have At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
* ECOG score of 0 ~ 2;
* Adequate bone marrow, hepatic and renal and coagulation function;
* Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
* Voluntarily participated in this study, signed the informed

Exclusion Criteria:

* Subjects who have received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc within 2 weeks before RT-01 administration;
* Subjects who have participate in another interventional study within 4 weeks before RT-01 administration;
* Subjects who have had major surgery within 4 weeks before RT-01 administration.
* Patients in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days before RT-01 administration, but currently or previously treated with any of the following steroid regimens, were included: Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption; Prophylactic short-term use of corticosteroids;
* Subjects who have participate in another oncolytic virus study within 8 weeks before RT-01 administration;
* Subjects received live vaccines within 7 days before RT-01 administration;
* Subjects received Antiviral drugs within 2 weeks, long-acting interferon within 4 weeks before RT-01 administration;
* Subjects with adverse reactions caused by previous anti-tumor treatment not recovered to (CTCAE 5.0) grade 1 (except alopecia);
* Subjects who have uncontrolled active infection;
* Subjects with known positive history of human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS);
* Subjects who have active hepatitis;
* Subjects who have serious cardiovascular system disorders history;
* Subjects with active autoimmune diseases or history of autoimmune diseases that may relapse;
* Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator;
* Subjects in other conditions that are considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.
To evaluate the antitumor activity | Up to 2 years
  To assessed per RECIST and iRECIST
The changes of the immunoreactivity during treatment. | Up to 28 days
  Peripheral blood T lymphocyte subtype
To evaluate the immunogenicity of RT-01 | Up to 28 days
  Antiviral antibody
To evaluate the viral shedding of RT-01 | Up to 24 Weeks
  Viral RNA
The Cmax of Viral RNA | Up to 24 Weeks
  The maximum RNA peak concentration
The Tmax of Viral RNA | Up to 24 Weeks
  The time of maximum RNA peak concentration

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No